CLINICAL TRIAL: NCT03525860
Title: The Feasibility of Acupuncture Treatment in the Post-Operative Cardio-Thoracic Setting for Arrhythmias in Patients Undergoing Open Heart Surgery- A Pilot Study
Brief Title: Acupuncture Treatment for Patients Who Develop Arrhythmias in the Post-Operative Cardio-Thoracic Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-006095
Record Dates: First submitted 2018-04-26; First posted 2018-05-16 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Post-Operative Atrial Fibrillation; Acupuncture Therapy
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture Treatment (Experimental): 20 subjects will be treated with standard of care and acupuncture.
  Will complete Symptom and Pain questionnaire (VAS) and a Was It Worth It (WIWI) questionnaire each day of study participation (3 days).
  Interventions: Procedure: Acupuncture
- No Intervention (No Intervention): 20 subjects will be treated with standard of care only.
  Will complete Symptom and Pain questionnaire (VAS) each day of study participation (3 days).

INTERVENTIONS:
Procedure: Acupuncture — The subject is placed in the selected position (lying down or sitting), based on their comfort level. The areas to be needled are prepped with an alcohol swab. Mandatory standards and safety guidelines for acupuncture will be followed.
  The acupuncture treatment protocol will be based on Traditional Chinese Medicine (TCM) theory. The TCM treatment strategy is designed to Benefit the Heart, Tonify Heart Qi and Blood, Calm and Sedate Cardiac Excitability and Regulate the Qi. Current literature supports the use of selected acupuncture points as possibly beneficial in regulating the autonomic nervous system, modulating Heart Rate Variability (HRV), relieving chest pain, and reducing arrhythmias.
  11 sterile, single use, disposable needles will be placed one by one until all needles are in place.
  Needles remain in place for additional 20 minutes or so as the patient remains in the selected position
  .
  Arms: Acupuncture Treatment

SUMMARY:
A feasibility study on the provision of acupuncture treatment in the hospital to 20 patients who have undergone open heart surgery procedures. The acupuncture treatments may begin as early as postoperative Day 2.

DETAILED DESCRIPTION:
Primary Aim • Evaluate the feasibility of providing acupuncture in the hospital setting for 20 patients undergoing open heart surgery and subsequently develop arrhythmias.

Secondary Aims

• Evaluate the short-term effect of acupuncture including the effects on patient's arrhythmias, stress, anxiety, and pain measured by Electrocardiogram monitoring and Electrocardiography, VAS scores, and WIWI questionnaire for the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have undergone CABG and/or cardiac valve operations.
2. Patients developing postoperative atrial fibrillation, and documented by ECG prior to acupuncture intervention, and treated with the common anti arrhythmic treatment of the department.
3. Patients moving to the step-down unit on postoperative day 2 or later.
4. Ability to provide informed consent.
5. Ability to speak English and complete all aspects of this trial.
6. At least 18 years of age.

Exclusion Criteria:

1. Patients with any other cardiac or non-cardiac concomitant procedures.
2. Patients with suspected sternal wound infection and/or with prolonged sternal wound dressing and wound- Vac-system application or open chest wound.
3. Patients with abnormal postoperative track staying in the intensive care unit for any clinical reason or hemodynamic compromise.
4. Patients with platelet count <50,000
5. Patients in a severe immunocompromised state.
6. Pregnant women. All patients who meet the criteria will have their medical records reviewed to ensure they are not pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
Acupuncture treatment in the hospital setting | 3 days post surgery
  The number of patients that complete acupuncture treatment in the hospital setting for patients having undergone heart surgery.

SECONDARY OUTCOMES:
Number of patients with recurrent atrial fibrillation | 3 consecutive days post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Chaim Leker Locker, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials